CLINICAL TRIAL: NCT03761433
Title: the Prediction of Postoperative Pain With Surgical Incision Stimulation in the Patients Undergoing Gastrectomy
Brief Title: Intraoperative Nociception and Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC2018-11-118
Record Dates: First submitted 2018-11-27; First posted 2018-12-03 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative; Nociceptive Pain; Analgesics
MeSH Terms: conditions — Pain, Postoperative; Nociceptive Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPI group: All patients who received the liver resection surgery will receive surgical pleth index
  Interventions: Device: SPI group

INTERVENTIONS:
Device: SPI group — All patients applied surgical pleth index at the time of surgical incision, under End tidal Sevoflurane 3%

SUMMARY:
If the individual patient's pain is assessed and the amount of analgesic needed after surgery is predicted, appropriate injection of pain control and excessive injection of narcotic analgesic can be prevented. Therefore, investigators try to evaluate the relation intraoperative nociception response with postoperative pain score.

In similar anesthetic depth(End tidal sevoflurane 3%) , changes of surgical pleth index values for stimulus of skin incision are thought to reflect the individual nociception characteristics.

DETAILED DESCRIPTION:
Patients who undergoing upper abdominal laparotomy surgery usually experience severe postoperative pain. Previous studies were reported that preoperative pain, young age, high-dose remifentanil, and depression were associated with severe postoperative pain.

However, anesthesia-related studies were either retrospective studies or injected with anesthetic agents in excess of clinical doses to differentiate between groups. There is no objective indicator for prediction severe postoperative pain.The purpose of this study was to investigate the relationship between intraoperative pain response and postoperative pain on standardized surveillance devices.

To maintain the depth of anesthesia, an EEG monitoring device bispectral index (BIS) is used. Also, surgical pleth index (SPI, GE healthcare, Freiburg, Germany) is a noninvasive pain-analgesia balance monitoring device that is commercially available to evaluate the state of pain during general anesthesia. SPI = 100- (0.3 * heart beat interval + 0.7 * photoplethysmographic pulse wave amplitude) is automatically and continuously calculated from the waveform of peripheral oxygen saturation.

In similar anesthetic depth(End tidal sevoflurane 3%) , changes of SPI values for stimulus of skin incision are thought to reflect the individual nociception characteristics. The investigators hypothesized the higher analgesics consumption can predict with high SPI response following incisional stimuli.

Thus, investigators try to evaluate the comparison of two groups ( high fentanyl consumption group vs. low fentanyl consumption group) with intraoperative SPI value (incision and before aurosal) and hemodynamic parameters under End tidal sevoflurane 3%(anesthesia depth, hemodynamically stable and appropriate anesthetic depth based on previous studies were confirmed at the time of skin incision). And the characteristics and emotional status of patients in two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

-undergoing laparotomy gastrectomy

Exclusion Criteria:

* cardiac arrythmia
* allergic history for drugs
* renal failure (Cr> 1.5 mg/dl)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the 20-80 year old patients who undergoing lapatotomy gastrectomy at samsung medical center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
The requirement of postoperative analgesics for postoperative 24 hours | postoperative 24 hour
  The requirement of postoperative analgesics for postoperative 24 hours (opioid conversion to fentanyl dose mcg)
The immediate postoperative pain score | postoperative 24 hour
  The numeric rating pain score, no pain=0 ~ worst pain=10
intraoperative nociception score (surgical pleth index) | intraoperative at the time of skin incision
  under End tidal sevoflurane 3%, surgical pleth index score following surgical incision

SECONDARY OUTCOMES:
The correlation of requirement of summed postoperative analgesics and intraoperative nociception score | postoperative 1 hour
  The consumption of analgesics (opioid conversion to fentanyl dose mcg) and intraoperative surgical pleth index value
The correlation of highest postoperative pain score and intraoperative nociception score | postoperative 1 hour
  The postoperative pain score (numeric rating pain score, no pain=0~ worst pain=10)and intraoperative surgical pleth index score

OTHER OUTCOMES:
The expectation of postoperative pain | The day before surgery
  The postoperative pain score (numeric rating pain score, no pain=0~ worst pain=10)
The expectation of analgesics consumption | The day before surgery
  less than average, average, more than average

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robertson TC, Hall K, Bear S, Thompson KJ, Kuwada T, Gersin KS. Transversus abdominis block utilizing liposomal bupivacaine as a non-opioid analgesic for postoperative pain management. Surg Endosc. 2019 Aug;33(8):2657-2662. doi: 10.1007/s00464-018-6543-z. Epub 2018 Nov 2. PMID 30390161
- [Background] Schreiber KL, Martel MO, Shnol H, Shaffer JR, Greco C, Viray N, Taylor LN, McLaughlin M, Brufsky A, Ahrendt G, Bovbjerg D, Edwards RR, Belfer I. Persistent pain in postmastectomy patients: comparison of psychophysical, medical, surgical, and psychosocial characteristics between patients with and without pain. Pain. 2013 May;154(5):660-668. doi: 10.1016/j.pain.2012.11.015. Epub 2012 Dec 5. PMID 23290256
- [Background] Ledowski T, Burke J, Hruby J. Surgical pleth index: prediction of postoperative pain and influence of arousal. Br J Anaesth. 2016 Sep;117(3):371-4. doi: 10.1093/bja/aew226. PMID 27543532
- [Background] Baron-Stefaniak J, Gotz V, Allhutter A, Schiefer J, Hamp T, Faybik P, Berlakovich G, Baron DM, Plochl W. Patients Undergoing Orthotopic Liver Transplantation Require Lower Concentrations of the Volatile Anesthetic Sevoflurane. Anesth Analg. 2017 Sep;125(3):783-789. doi: 10.1213/ANE.0000000000002250. PMID 28678075